CLINICAL TRIAL: NCT00180687
Title: Prospective Double Blind Randomized Controlled Trial of the Use of Intraperitoneal Nebulised Local Anaesthetic
Brief Title: Clinical Trial of the Use of Intraperitoneal Local Anaesthetic
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Principal Investigator, Nawar Alkhamesi, Clinical Research Fellow, Imperial College London
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 02.CD/218E; Dr. David Peck (Other: Imperial College London); Prof. Sir Ara Darzi (Other: Imperial College London)
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Results first posted 2015-09-15 (Estimated); Last update posted 2015-09-15 (Estimated); Status verified 2015-08

CONDITIONS: Pain, Postoperative
Keywords: Pain; Nebulisation; Cholecystectomy; Laparoscopic; Bupivacaine; Local Anaesthetic
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Bupivacaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Control (Sham Comparator): No intraperitoneal therapeutics (No nebulised Bupivacaine)
  Interventions: Other: No Intraperitoneal Therapeutics
- IP Aerosolized Normal Saline (Placebo Comparator): Intraperitoneal nebulised 10mls. Normal Saline (No nebulised Bupivacaine)
  Interventions: Drug: Normal Saline
- Nebulised Bupivacaine intraperitoneally (Experimental): Intraperitoneal Nebulised 10mls. Bupivacaione (Marcaine)
  Interventions: Drug: Nebulised Bupivacaine intraperitoneally
- Injected Bupivacaine intraperitoneally (Active Comparator): Intraperitoeal Injected 10 mls.Bupivacaine (Marcaine) (No nebulised Bupivacaine)
  Interventions: Drug: Injected Bupivacaine intraperitoneally

INTERVENTIONS:
Drug: Nebulised Bupivacaine intraperitoneally — Nebulised Marcaine (Bupivacaine)
  Other Names: Marcaine
  Arms: Nebulised Bupivacaine intraperitoneally
Drug: Normal Saline — Nebulised Normal Saline
  Other Names: 0.9 % Normal Saline
  Arms: IP Aerosolized Normal Saline
Drug: Injected Bupivacaine intraperitoneally — Injected Marcaine directly into the peritoneal cavity
  Other Names: Marcaine
  Arms: Injected Bupivacaine intraperitoneally
Other: No Intraperitoneal Therapeutics — No Intraperitoneal Therapeutics given
  Arms: Control

SUMMARY:
Patients undergoing keyhole gall bladder removal will be divided into 3 groups, one control, one will have local anaesthetic and the third will have normal saline nebulised into their abdomen before closure of the wounds to reduce postoperative pain. These medications will be given on top of the standard pain management protocol.

DETAILED DESCRIPTION:
Pain post laparoscopic procedures can be divided into access related, operation site and distension related. The access type can be attenuated by the use of sub dermal infiltration of local anaesthetic and rarely causes significant discomfort. It has been advocated that placement of a peritoneal gas drain significantly reduces postoperative pain particularly referred to the shoulder tip. Realistically, however, if attention is paid to expelling the residual gas at the end of the procedure this complication is rarely problematic. Operative site pain however is more difficult to manage. In limited gynaecological procedures it has been shown that local installation of local anaesthetic decreased the analgesic requirement of patients post operatively. These observations would not be as transferable to more extensive colorectal or solid organ surgery as the amount of local anaesthesia required would be toxic to the patient. Use of the nebuliser, however maybe able to alleviate pain by efficiently using the dosage required.

This is a prospective randomised double blind trial. Sixty patients will be allocated randomly between three groups, 20 patients in each group:

1. Control group
2. Nebulised intraperitoneal local anaesthetic (Bupivacaine 0.25%, 3mg/Kg)
3. Nebulised intraperitoneal normal saline Ward staff will be blinded to which group the patients are in. All patients undergoing laparoscopic cholecystectomy who have given written, informed consent are eligible for inclusion. Patients with local anaesthetics allergy and patients whom pain evaluation is considered unreliable due to chronic opiate use or neurological diseases are excluded.

No pre-medication is to be given and a standardised anaesthetic technique is to be employed for all patients.

Standard 4 ports technique for laparoscopic cholecystectomy will be used with intraperitoneal pressure between 12-14 mmHg. This will be achieved using CO2 as the insufflation gas.

The local anaesthetic (approximately 10mls) will be delivered via a fine sterile catheter that will be inserted via the epigastric port under direct vision at the end of the procedure. Afterward the pneumoperitoneum will be deflated and the wound will be closed and subcutaneous local anaesthetic will be injected in and around the wounds.

Postoperatively, all the patients will have PCA as the main analgesia supported by NSAIDs unless contraindicated. Patients will eat and drink as desired and drips will be taken as soon as it is safe to do so.

Postoperative pain scoring will be stared in recovery and continue on the wards using the visual analogue scale.

ELIGIBILITY:
Inclusion Criteria:

* All they patients undergoing laparoscopic cholecystectomy will be included.

Exclusion Criteria:

* Patients with local anaesthetic allergy, patients on chronic opiate medication or those with neurological diseases that make pain evaluation unreliable will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2004-10; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nawar A Alkhamesi, MD, PhD, Principal Investigator — Imperial College London
Locations (1):
- St. Mary's Hospital, London, United Kingdom

REFERENCES:
- [Result] Alkhamesi NA, Peck DH, Lomax D, Darzi AW. Intraperitoneal aerosolization of bupivacaine reduces postoperative pain in laparoscopic surgery: a randomized prospective controlled double-blinded clinical trial. Surg Endosc. 2007 Apr;21(4):602-6. doi: 10.1007/s00464-006-9087-6. Epub 2006 Dec 16. PMID 17180268

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | IP Aerosolized Normal Saline | Nebulised Bupivacaine Intraperitoneally | Injected Bupivacaine Intraperitoneally
Started | 20 | 20 | 20 | 20
Completed | 20 | 20 | 20 | 20
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | IP Aerosolized Normal Saline | Nebulised Bupivacaine Intraperitoneally | Injected Bupivacaine Intraperitoneally | Total
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 80
Age, Continuous [Mean (Full Range); unit: Years] | 47.65 [25 to 75] | 47.65 [26 to 74] | 51.60 [25 to 83] | 48.70 [34 to 79] | 49 [25 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 18 | 17 | 18 | 69
  Male | 4 | 2 | 3 | 2 | 11
Region of Enrollment [Number; unit: participants]
  United Kingdom | 20 | 20 | 20 | 20 | 80

OUTCOME MEASURES:

1. Primary Outcome: Reduction in Postoperative Pain
Description: Postoperative pain was measured using Pain scale 0-10 (0 = No Pain, 10 = Maximum pain). A trained nursing staff will ask the patient about his / her pain and document that correctly in the chart. The staff will also document if the patient requires any analgesia, the type and the dose.
Time Frame: 0 hours, 6 hours, 12 hours, 24 hours
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Control | IP Aerosolized Normal Saline | Nebulised Bupivacaine Intraperitoneally | Injected Bupivacaine Intraperitoneally
Number analyzed (Participants) | 20 | 20 | 20 | 20
units on a scale
  Pain in Recovery (0 Hours) | 9.2 [3 to 10] | 10 [10 to 10] | 3.3 [1 to 10] | 9.3 [5 to 10]
  Pain at 6 hours | 8.2 [5 to 10] | 8.1 [4 to 10] | 0.7 [0 to 3] | 7.2 [4 to 10]
  Pain at 12 hours | 7.9 [3 to 10] | 8 [4 to 10] | 0.6 [0 to 3] | 6.7 [4 to 10]
  Pain at 24 hours | 6.1 [4 to 10] | 6.2 [2 to 10] | 0.5 [0 to 3] | 5.6 [3 to 8]

2. Secondary Outcome: Number of Vomiting / Nausea Episodes
Description: Nausea and vomiting are known adverse effect of opioids usage. By reducing the use of opioids we can reduce or abolish these side effect which will enhance early patient recovery and discharge and reduce hospital cost. We will measure the number of episodes when the patient suffers from these side effect and correlate them with opioids use.
Time Frame: 24 hours
Measure: Mean (Full Range); unit: Number of vomitting / Nausea episodes
Arm/Group | Control | IP Aerosolized Normal Saline | Nebulised Bupivacaine Intraperitoneally | Injected Bupivacaine Intraperitoneally
Number analyzed (Participants) | 20 | 20 | 20 | 20
Number of vomitting / Nausea episodes | 7.1 [5 to 9] | 7.1 [3 to 8] | 2 [0 to 4] | 6.8 [2 to 9]

3. Secondary Outcome: Hours Needed for Safe Mobilization
Description: Drowsiness and delayed mobilization are known adverse effect of opioids usage. By reducing the use of opioids we can reduce or abolish these side effect which will enhance early patient recovery and discharge and reduce hospital cost. We will measure how many hours will take the patient to mobilize freely and safely and correlate them with opioids use.
Time Frame: 24 Hours
Measure: Mean (Full Range); unit: Hours needed for safe mobilization
Arm/Group | Control | IP Aerosolized Normal Saline | Nebulised Bupivacaine Intraperitoneally | Injected Bupivacaine Intraperitoneally
Number analyzed (Participants) | 20 | 20 | 20 | 20
Hours needed for safe mobilization | 6.7 [4 to 10] | 6.5 [4 to 11] | 3 [2 to 4] | 6.4 [3 to 9]

4. Secondary Outcome: Postoperative Morphine Use
Description: The reduction in cost comes from reducing the use of opioid which requires nursing supervision and also special pump to be delivered as in the cases of patient controlled analgesia. With that reduction, there will be a reduction in opioid related adverse events that mandate medical or nursing attention and prolong hospitalization, these adverse events include nausea and vomiting, delay mobilization due to drowsiness and alter mental status caused by opioid usage. For these reasons we are collecting data related to these adverse events
Time Frame: 24 Hoiurs
Measure: Mean (Full Range); unit: mg
Arm/Group | Control | IP Aerosolized Normal Saline | Nebulised Bupivacaine Intraperitoneally | Injected Bupivacaine Intraperitoneally
Number analyzed (Participants) | 20 | 20 | 20 | 20
mg | 25.9 [10 to 45] | 26.3 [10 to 50] | 1 [0 to 10] | 16.7 [8 to 30]

ADVERSE EVENTS:
Time Frame: 24 Hours
Description: Nausea and Vomiting
Arm/Group | Control | IP Aerosolized Normal Saline | Nebulised Bupivacaine Intraperitoneally | Injected Bupivacaine Intraperitoneally
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 5/20 | 5/20 | 1/20 | 5/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=20) | IP Aerosolized Normal Saline (N=20) | Nebulised Bupivacaine Intraperitoneally (N=20) | Injected Bupivacaine Intraperitoneally (N=20)
Nausea and Vomiting (Gastrointestinal disorders) | 5 (9) | 5 (8) | 1 (4) | 5 (9) — Number of Nausea / vomiting episodes recorded in patient's chart

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes